CLINICAL TRIAL: NCT06652425
Title: Acute Effects of Cold Exposure on Cardiovascular System and Potential Mechanism in Healthy Young Adults: A Randomized Controlled Study
Brief Title: Acute Effects of Cold Exposure on Cardiovascular System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Renjie Chen, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#2024-10-1167
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular System
Keywords: Low temperature; Randomized controlled trial; Cardiovascular system
MeSH Terms: interventions — Cold Temperature; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low temperature (15°C) group (Experimental): Subjects in exposure group will be exposed to low temperature (15°C) for about 2 hours in a chamber.
  Interventions: Other: Low temperature (15°C) group
- Moderate temperature (22°C) group (Experimental): Subjects in exposure group will be exposed to moderate temperature (22°C) for about 2 hours in a chamber.
  Interventions: Other: Moderate temperature (22°C) group

INTERVENTIONS:
Other: Low temperature (15°C) group — The exposure group will be exposed to low temperature (15°C) in a chamber for about 2 hours, resting during the whole periods.
  Arms: Low temperature (15°C) group
Other: Moderate temperature (22°C) group — The exposure group will be exposed to thermoneutral temperature (22°C) in a chamber for about 2 hours, resting during the whole periods.
  Arms: Moderate temperature (22°C) group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aim to assess the acute effects of low temperature exposure on cardiovascular system and the underlying mechanisms.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled human exposure crossover study among about 40 healthy young adults in Shanghai, China. Each subject will be exposed twice: once to the low temperature (15°C) and once to the moderate temperature (22°C) in a chamber for about 2 hours. During the exposure session, each subject will be requested to rest. Health examinations will be conducted at baseline immediately prior to exposure, during the period of exposure, and after exposure. Health examinations include blood pressure tests and Holter monitoring. Investigators plan to collect blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Body mass index > 18.5 and ≤ 28;
* Right-handed;
* Receiving or having received higher education;
* With the ability to read and understand Chinese smoothly.

Exclusion Criteria:

* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory diseases, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects who have a history of major surgery due to cardiovascular, cerebrovascular, respiratory, or neurological diseases;
* Subjects with neurologic disorders, such as stroke, traumatic brain injury, epilepsy, and schizophrenia;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Subjects with color vision disabilities.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Blood pressure will be examined before exposure and immediately after the exposure session
  The changes of systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured.
SDNN (standard deviation of NN intervals) | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure heart rate variability (HRV) parameter SDNN
SDANN (standard deviation of the averages of RR intervals) | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure heart rate variability parameter SDANN
rMSSD (root mean square of successive differences) | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure heart rate variability (HRV) parameter rMSSD
pNN50 (Percentage of differences between adjacent RR intervals greater than 50 ms) | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure heart rate variability (HRV) parameter pNN50
Frequency domain measures: low frequency (LF), high frequency (HF), and LF/HF ratio | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure frequency domain parameters of heart rate variability (HRV)

SECONDARY OUTCOMES:
Changes of scores of symptoms questionnaires | The questionnaires will be conducted before exposure and immediately after the exposure
  The changes of scores of respiratory and cardiovascular symptoms questionnaires both the total and each symptom specified
Changes of skin temperature | Skin temperature will be examined during the 2-hour exposure session
  The changes of wrist skin temperature will be measured

OTHER OUTCOMES:
Differences in metabolic profiling detected in blood between the two exposures | 1 hour after the exposure session
  The differential metabolic profiling in blood related to high temperature exposurewill be detected by maspectrometrybased non-targeted metabolomics.
Differences in protein levels detected in blood between the two exposures | 1 hour after the exposure session
  The differentially expressed proteins in blood related to high temperature exposure will be detected by non-targeted proteomics.
Differences in RNA expression levels detected in serum transcriptomics between the two exposures | 1 hour after the exposure session
  Illumina-based transcriptomics is non-targeted. The study is to find the differentially expressed exosome RNA in serum after low temperature exposure
Differences in DNA methylation levels detected in whole-blood between the two exposures | 1 hour after the exposure session
  Genome-wide DNA methylation in whole-blood were detected. The study is to identify differential CpG loci after low temperature exposure
Changes of the scores of thermal sensation questionnaires | The questionnaires will be conducted before exposure and immediately after the exposure session
  Changes of scores of thermal sensation questionnaires which ranged from -5 to 5. Zero score refers to the thermal comfort sensation. Higher scores refer to more uncomfortable sensations of hot. Lower scores refer to more uncomfortable sensations of cold.
Change in serum CRP concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of C reactive protein in blood.
Change in serum APOA1 concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of APOA1 in blood will be measured.
Change in serum APOB concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of APOB in blood will be measured.
Change in serum Cholesterol concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of Cholesterol in blood will be measured.
Change in serum Glucose concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of Glucose in blood will be measured.
Change in serum HDL concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of HDL in blood will be measured.
Change in serum Insulin concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of Insulin in blood will be measured.
Change in serum LDL concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of LDL in blood will be measured.
Change in serum LPa concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of LPa in blood will be measured.
Change in serum TG concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of TG in blood will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT06652425/Prot_SAP_000.pdf